# Georgia State University Informed Consent

<u>Title:</u> Panthers4Life: A pilot randomized controlled trial to test the efficacy of a brief intervention among high-risk college students

Principal Investigator: Amanda K. Gilmore, PhD

**Sponsor:** Substance Abuse and Mental Health Services Administration

## **Introduction and Key Information**

- You are invited to take part in a research study. It is up to you to decide if you would like to take part in the study. You may stop at any time.
- The purpose of this study is to learn if a program for college students is helpful. The program is about alcohol use among college students.
- You will be asked to answer questions to see if you are eligible. If you are eligible, you will complete a 15-minute online survey about college students' health and behaviors. You may be randomly selected to complete a 15-minute online program about alcohol use. You will be emailed a link 3 months later to complete another 15-minute online survey.
- Your role in this study will last between 30-45 minutes and will span over the course of 3 months.
- If you do not want to be in this study, your other choice is to not consent and not participate in the study.

#### **Purpose**

The purpose of this study is to learn if a program for college students is helpful. You are invited to take part in this research study because you are a college student aged 18-25. A total of 400 college students from Georgia State University will be asked to participate in this study.

## **Procedures**

If you decide to take part, you will:

- Answer questions about your race, ethnicity, sexual orientation, gender identity, sex at birth, and alcohol use to see if you are eligible for the study.
- If you are eligible and want to be in the study, you will complete a 15-minute online survey about college students' health and behaviors. This includes alcohol use, sexual experiences, stress, and post-traumatic stress disorder.
- After answering questions, you will be randomly redirected to take the online program or not (random like a coin flip). The online program takes about 15 minutes, and you will read

Version Date: 6-21-2023

- information and answer interactive questions about alcohol use. If you do not receive the program, you will be directed to a website with resources for substance use and mental health.
- Then, you will be emailed a link 3 months later and asked to complete an online survey about college students' health and behaviors.
- Today's activities will last between 15-30 minutes if you are eligible for the study (but only 5 minutes if you are not eligible). The 3-month follow-up survey will take another 15 minutes.

#### **Future Research**

Researchers will remove information that may identify you and may use your data for future research. If we do this, we will not ask for any additional consent from you.

#### Risks

You will not have any more risks than you would in a normal day of life. No injury is expected from this study. If you believe you have been harmed, contact the research team as soon as possible. Georgia State University and the research team have not set aside funds to compensate for any injury.

#### **Benefits**

This study is not designed to benefit you personally, but if you get the program, it might help your health and give you more information about your alcohol use. If you do not get the program, the resources provided may have health benefits if utilized. Overall, we hope to gain information from the study to help make programs better for college students like you.

# **Alternatives**

The alternative to taking part in this study is to not take part in the study.

## Compensation

If you are eligible to participate and enrolled in this study, you will be paid \$30 for completing all procedures in this study. You will be paid \$15 for the baseline survey and \$15 for the 3-month follow-up survey.

## **Voluntary Participation and Withdrawal**

You do not have to be in this study. If you decide to be in the study and change your mind, you have the right to drop out at any time. You may skip questions or stop participating at any time. This will not cause you to lose any benefits to which you are otherwise entitled.

# Confidentiality

We will keep your records private to the extent allowed by law. The following people and entities will have access to the information you provide:

- Dr. Amanda Gilmore and her research team
- Georgia State University Institutional Review Board
- Office for Human Research Protection (OHRP)

Version Date: 6-21-2023

• Substance Abuse and Mental Health Services Administration

We will use a study number rather than your name on study records. The information you provide will be stored in a locked cabinet and/or on password- and firewall-protected computers. Data sent over the internet may not be secure. All data collection is completed on websites with encryption to protect your identity. Your study number will be stored separately from the data to protect privacy. When we present or publish the results of this study, we will not use your name or other information that may identify you.

# **Contact Information**

Contact Amanda K. Gilmore, PhD at <a href="mailto:panthers4life@gsu.edu">panthers4life@gsu.edu</a>

- If you have questions about the study or your part in it
- If you have questions, concerns, or complaints about the study
- If you think you have been harmed by the study

The IRB at Georgia State University reviews all research that involves human participants. You can contact the IRB if you would like to speak to someone who is not involved directly with the study. You can contact the IRB for questions, concerns, problems, information, input, or questions about your rights as a research participant. Contact the IRB at 404-413-3500 or irb@gsu.edu.

| You can print or save a copy of this form for your records. |
|-----------------------------------------------------------------------|
| Please indicate below whether you agree to participate in this study. |
| _ I agree to participate, continue to study |
| _ I do not agree to participate, do not continue to study |